CLINICAL TRIAL: NCT05229965
Title: Paracetamol Vs Paracetamol-Caffeine Association Vs Paracetamol-Codeine Association in the Management of Post Traumatic Pain in Emergencies
Brief Title: Paracetamol Vs Caffeine Vs Codeine in the Management of Post Traumatic Pain in Emergencies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, PROFESSOR, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Codeine-Cafeine-Paracetamol
Record Dates: First submitted 2021-12-08; First posted 2022-02-08 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Acute Pain Due to Trauma
Keywords: acute pain; trauma; paracetamol; codeine; cafeine
MeSH Terms: conditions — Acute Pain; Wounds and Injuries | interventions — Acetaminophen; acetaminophen, codeine drug combination

STUDY DESIGN:
Who Masked: Participant
Masking Description: study medications consists of a randomly sequence generated numbers.
  patients and the research associate who collected the outcome data are blinded from the study group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paracétamol Group (Active Comparator): In each study population, the patient will be assigned to one of three treatments (Paracetamol Group or Paracetamol Codéine Group or Paracétamol Caféine Group) .
  In Paracetamol group , the patients will receive a pill containing 1000 mg of paracetamol 3 times a day for 7 days .
  Paracétamol 1000 mg : 1 pill *3 / day
  Interventions: Drug: Paracetamol
- Paracétamol Codéine Group (Active Comparator): In each study population, the patient will be assigned to one of three treatments (Paracetamol Group or Paracetamol Codéine Group or Paracetamol Caféine Group) .
  In Paracetamol codéine group , the patients will receive a pill containing an association of paracetamol and codéine ( 500mg / 30mg ) 3 times a day for 7 days .
  -Association of Paracétamol and Codéine ( 500mg / 30 mg) : 1 pill *2 /day
  Interventions: Drug: Paracetamol Codeine
- Paracétamol Caféine Group (Active Comparator): In each study population, the patient will be assigned to one of three treatments (Paracetamol Group or Paracetamol Codéine Group or Paracetamol Caféine Group) .
  In Paracetamol caféine group , the patients will receive a pill containing an association of paracetamol and caféine ( 500mg / 65 mg ) 3 times a day for 7 days .
  -Association of Paracétamol and Caféine ( 500mg / 65 mg) : 1 pill *3 /day
  Interventions: Drug: Paracetamol caféine

INTERVENTIONS:
Drug: Paracetamol — 21 pills will be provided with a preconised dose of 1 pill 3 times per day over 7 days period
  Other Names: 1000mg
  Arms: Paracétamol Group
Drug: Paracetamol Codeine — 14 pills will be provided with a preconised dose of 1 pill 2 times per day over 7 days period
  Other Names: 500mg/ 30mg
  Arms: Paracétamol Codéine Group
Drug: Paracetamol caféine — 21 pills will be provided with a preconised dose of 1 pill 3 times per day over 7 days period
  Other Names: 500mg/ 65mg
  Arms: Paracétamol Caféine Group

SUMMARY:
The purpose of this study is to:

Compare the effect of paracetamol alone against Paracetamol+Codeine association against the association of paracetamol + Cafeine in the treatment of post-traumatic acute pain of the limbs.

DETAILED DESCRIPTION:
At admission to the emergency department, patients with acute post-traumatic pain will be included, regardless of their initial NRS .These patients will receive the necessary care for their injury (icing, reduction, immobilization, local care, sutures), then went home with a medical prescription and an outpatient appointment .

At discharge and after obtaining their signed consent . All patients included will be randomized according to a numerical randomization table ( assigned in a 1:1:1 ratio) into 3 groups ( As a treatment for their post traumatic pain at discharge for 7 days ) :

* Group 1: Paracetamol group who will receive paracetamol ( 1000 mg) : one pill 3 times a day for 7 days .
* Group 2: Paracetamol-codeine group who will receive an association of 500 mg of Paracetamol and 30 mg of codeine : one pill twice a day for 7 days .
* Group 3: Paracetamol-cafeine group who will receive an association of 500 mg of Paracetamol and 65 mg of cafeine : one pill 3 times a day for 7 days .

For all patients included in the study, demographic and clinical data will be collected by the physician or investigator and recorded on a pre-established form.

The demographic data recorded on each patient's chart were as follows: Age, sex, origin and personal pathological history:

* Hypertension.
* Diabetes.
* Respiratory insufficiency.
* Renal insufficiency.
* Liver failure.
* Allergy.

And a Clinical examination data:

* Pain intensity (NRS).
* Mechanism of trauma and site of injury.
* Other physical examination data: systolic blood pressure (SBP), heart rate (HR) and temperature.
* Nature of traumatic injury.
* Final diagnosis
* Injury Severity Score (ISS).
* NRS at discharge (at rest and on movement).

Patients included will be assessed at Day 1 , Day 2 , Day 3 and Day 7 after discharge from the emergency department by a telephone call. This evaluation will include :

* NRS at rest and during movement
* Secondary use of another analgesic.
* Patient satisfaction assessed by Likert scale, with 3 responses:

  * Satisfied
  * Moderately satisfied
  * Not satisfied
* Side effects: epigastralgia, dizziness, somnolence, headache, nausea and/or vomiting, insomnia, constipation, palpitation, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age :18 years or older
* Patients presented to the emergency department with acute post-traumatic pain and residual pain at rest and/or on movement with a numerical pain rating scale (NRS) > 3/10 on discharge.
* They all signed a written consent form.

Exclusion criteria:

* Self-mutilation
* Severe acute trauma that may require hospitalization
* Open or complicated fracture requiring surgical management
* Regular use of analgesics
* Any known allergy to paracetamol, caffeine or codeine
* Asthma and acute/chronic respiratory insufficiency
* Severe renal insufficiency (creatinine Cl<30 ml/min)
* Pregnant/lactating women
* Hepatic cirrhosis.
* Refusal, incapacity or difficulties to consent or to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Delta Numerical Rating Scale (NRS) ( From 0 to 10 ) | 7 days from discharge
  Treatment success is defined by the percentage of patients with a reduction in movement NRS at Day 7 discharge (Delta NRS ) ≥ 50% compared with NRS at emergency discharge. ( that mean a better outcome )
  Delta NRS ( in movement)=(NRS (at discharge )-NRS (day7))/(NRS (at discharge )) X 100 .

SECONDARY OUTCOMES:
Appearance of side effects | 7 days from discharge
  The appearance of side effects such as Drowsiness ,Decreased respiratory rate (<14 c / min), Cutaneous rash, Vomiting,Nausea,pruritus, Dizziness and Digestive hemorrhage.
Need for another analgesic medication or non-pharmacological analgesic intervention | 7 days from discharge
  The patient's need to add another analgesic medication or non-pharmacological analgesic intervention
Patient satisfaction assessed by Likert's verbal scale at 7 days | 7 days from discharge
  patient satisfaction assessed by Likert's verbal scale : with 3 responses:
  * Satisfied
  * Moderately satisfied
  * Not satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Principal Investigator — Monastir University Hospital, Monastir, Tunisia, 5000
Locations (1):
- Nouira Semir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No